CLINICAL TRIAL: NCT03306862
Title: A Randomized, Controlled, Cross-over Trial Examining the Effect of Peas in Soup on Post-prandial Glycaemic Response in Healthy Adults.
Brief Title: Effect of Peas in Soup on Blood Glucose Control
Acronym: PEA4
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government); University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Heather Blewett, Principal Investigator, St. Boniface Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: RRC/2017/1704; HS21196 (B2017:123) (Other: Biomedical Research Ethics Board, University of Manitoba)
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Post-prandial Glycaemia
Keywords: blood sugar; insulin; peas
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Whole yellow pea (Experimental): Soup containing 25g available carbohydrates from whole yellow peas. Intervention: Whole yellow pea soup
  Interventions: Dietary Supplement: Whole yellow pea soup
- Split yellow pea (Experimental): Soup containing 25g available carbohydrates from split yellow peas. Intervention: Split yellow pea soup
  Interventions: Dietary Supplement: Split yellow pea soup
- Potato (Placebo Comparator): Soup containing 25g available carbohydrates from potatoes. Intervention: Potato soup
  Interventions: Dietary Supplement: Potato soup

INTERVENTIONS:
Dietary Supplement: Whole yellow pea soup — Soup containing whole yellow peas
  Arms: Whole yellow pea
Dietary Supplement: Split yellow pea soup — Soup containing split yellow peas
  Arms: Split yellow pea
Dietary Supplement: Potato soup — Soup containing potatoes
  Arms: Potato

SUMMARY:
This study is part of a group of studies whose overall goal is to accurately define the physiochemical and structural effects of pea varieties and relate these to blood glucose attenuation in healthy human volunteers.

DETAILED DESCRIPTION:
A randomized, controlled, cross-over study designed to examine the post-prandial glycaemic response to peas in soup will be conducted at the I.H. Asper Clinical Research Institute in Winnipeg, Manitoba. Eligible participants who have provided consent will be asked to attend 3 clinic visits in a fasted state. Participants will be given soup containing peas at 2 visits and soup without peas at 1 visit. At each visit participants will provide 7 capillary blood samples via finger poke, 5 questionnaires about their appetite and a questionnaire about the acceptability of the products. Each visit will last approximately 2.5h and be separated by 3-14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy male or female, between the age of 18-40 years;
2. Body mass index (BMI) 18.5-30.0 kg/m2;
3. Habitually consume breakfast, lunch and dinner in the morning, mid-day and evening, respectively.
4. Willing to provide informed consent;
5. Willing/able to comply with the requirements of the study.

Exclusion Criteria:

1. Pregnant or lactating;
2. Medical history of diabetes mellitus, fasting blood glucose ≥6.1 mmol/L, HbA1c ≥6.0%, or use of insulin or oral medication to control blood sugar;
3. Medical history of cardiovascular disease;
4. Systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg;
5. Fasting plasma total cholesterol >7.8 mmol/L;
6. Fasting plasma HDL <0.9 mmol/L;
7. Fasting plasma LDL >5.0 mmol/L;
8. Fasting plasma triglycerides >2.3 mmol/L;
9. Major surgery within the last 3 months;
10. Medical history of inflammatory disease (ie. Systemic lupus erythematosis, rheumatoid arthritis, psoriasis) or use of any corticosteroid medications within 3 months;
11. Medical history of liver disease or liver dysfunction (defined as plasma AST or ALT ≥1.5 times the upper limit of normal (ULN));
12. Medical history of kidney disease or kidney dysfunction (defined as blood urea nitrogen and creatinine ≥ 1.8 times the ULN));
13. Presence of a gastrointestinal disorder, daily use of any stomach acid-lowering medications or laxatives (including fibre supplements) within the past month or antibiotic use within the past 6 weeks;
14. Active treatment for any type of cancer within 1 year prior to study start;
15. Shift worker (a system of employment where an individual's normal hours of work are in part, outside the period of normal working day; 6am and 8pm);
16. Smoking, use of tobacco or a nicotine replacement product (within the last 3 months);
17. Allergies to peas;
18. Aversion or unwillingness to eat study foods;
19. Consuming >4 servings of pulses per week;
20. Use of any prescription or non-prescription drug, herbal or nutritional supplement known to affect glycaemia or appetite;
21. Participation in another clinical trial, current or in the past 4 weeks;
22. Unstable body weight (defined as >5% change in 3 months) or actively participating in a weight loss program.
23. Other medical, psychiatric, or behavioral factors that in the judgment of the principal Investigator may interfere with study participation or the ability to follow the intervention protocol;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Post-prandial glucose | 120 min
  iAUC for glucose
Post-prandial insulin | 120 min
  iAUC for insulin

SECONDARY OUTCOMES:
Hunger | 120 min
  AUC using visual analog scales
Fullness | 120 min
  AUC using visual analog scales
Desire to eat | 120 min
  AUC using visual analog scales
Prospective consumption | 120 min
  AUC using visual analog scales

OTHER OUTCOMES:
Acceptability of soup color | 15 min
  Ratings on a scale of 1-9
Acceptability of soup aroma | 15 min
  Ratings on a scale of 1-9
Acceptability of soup flavor | 15 min
  Ratings on a scale of 1-9
Acceptability of soup texture | 15 min
  Ratings on a scale of 1-9
Frequency of eating soup | 15 min
  Ratings on a scale of 1-9
Gastrointestinal side effects | 24 h
  Incidence of gastrointestinal effects

CONTACTS AND LOCATIONS:
Overall Officials: Heather Blewett, PhD, Principal Investigator — Agriculture and Agri-Food Canada
Locations (1):
- I.H. Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From the time the data is collected until the manuscript is accepted for publication.
Access Criteria: Dan Ramdath, Sora Ludwig and Michel Aliani will have access to data necessary for manuscript preparation.

REFERENCES:
- [Background] Public Health Agency of Canada and the Canadian Institute for Health Information. Obesity in Canada: A joint report from the Public Health Agency of Canada and the Canadian institute for health information. Government of Canada; 2011.
- [Background] Public Health Authority of Canada. Diabetes in Canada: Facts and figures from a public health perspective. 2011.
- [Background] Sievenpiper JL, Kendall CW, Esfahani A, Wong JM, Carleton AJ, Jiang HY, Bazinet RP, Vidgen E, Jenkins DJ. Effect of non-oil-seed pulses on glycaemic control: a systematic review and meta-analysis of randomised controlled experimental trials in people with and without diabetes. Diabetologia. 2009 Aug;52(8):1479-95. doi: 10.1007/s00125-009-1395-7. Epub 2009 Jun 13. PMID 19526214
- [Background] Hamberg O, Rumessen JJ, Gudmand-Hoyer E. Blood glucose response to pea fiber: comparisons with sugar beet fiber and wheat bran. Am J Clin Nutr. 1989 Aug;50(2):324-8. doi: 10.1093/ajcn/50.2.324. PMID 2547300
- [Background] Marinangeli CP, Jones PJ. Chronic intake of fractionated yellow pea flour reduces postprandial energy expenditure and carbohydrate oxidation. J Med Food. 2011 Dec;14(12):1654-62. doi: 10.1089/jmf.2010.0255. PMID 22145774
- [Background] Smith CE, Mollard RC, Luhovyy BL, Anderson GH. The effect of yellow pea protein and fibre on short-term food intake, subjective appetite and glycaemic response in healthy young men. Br J Nutr. 2012 Aug;108 Suppl 1:S74-80. doi: 10.1017/S0007114512000700. PMID 22916818
- [Background] Jenkins DJ, Thorne MJ, Camelon K, Jenkins A, Rao AV, Taylor RH, Thompson LU, Kalmusky J, Reichert R, Francis T. Effect of processing on digestibility and the blood glucose response: a study of lentils. Am J Clin Nutr. 1982 Dec;36(6):1093-101. doi: 10.1093/ajcn/36.6.1093. PMID 6293296
- [Background] Li H, Song F, Xing J, Tsao R, Liu Z, Liu S. Screening and structural characterization of alpha-glucosidase inhibitors from hawthorn leaf flavonoids extract by ultrafiltration LC-DAD-MS(n) and SORI-CID FTICR MS. J Am Soc Mass Spectrom. 2009 Aug;20(8):1496-503. doi: 10.1016/j.jasms.2009.04.003. Epub 2009 Apr 14. PMID 19443236
- [Background] Habtemariam S. A-glucosidase inhibitory activity of kaempferol-3-O-rutinoside. Nat Prod Commun. 2011 Feb;6(2):201-3. PMID 21425674
- [Background] Ames N, Blewett H, Storsley J, Thandapilly SJ, Zahradka P, Taylor C. A double-blind randomised controlled trial testing the effect of a barley product containing varying amounts and types of fibre on the postprandial glucose response of healthy volunteers. Br J Nutr. 2015 May 14;113(9):1373-83. doi: 10.1017/S0007114515000367. Epub 2015 Apr 8. PMID 25850814
- [Background] Rabiee A, Magruder JT, Grant C, Salas-Carrillo R, Gillette A, DuBois J, Shannon RP, Andersen DK, Elahi D. Accuracy and reliability of the Nova StatStrip(R) glucose meter for real-time blood glucose determinations during glucose clamp studies. J Diabetes Sci Technol. 2010 Sep 1;4(5):1195-201. doi: 10.1177/193229681000400519. PMID 20920440